CLINICAL TRIAL: NCT01476111
Title: A Prospective, Exploratory Observational Study Evaluating Specific Biomarkers in Primary Invasive Breast Cancer and Their Modulation by Standard Neoadjuvant Therapy
Brief Title: Evaluation of Specific Biomarkers in Primary Invasive Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Study termination due to negative Phase III of another study product from same technology platform.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115400
Record Dates: First submitted 2011-11-10; First posted 2011-11-22 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-02

CONDITIONS: Neoplasms, Breast
Keywords: tumor antigens; observational; breast cancer; biomarkers; Neoadjuvant
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue

GROUPS / COHORTS (1):
- Group 1: Patients with primary invasive breast cancer

SUMMARY:
This study will examine specific biomarkers in primary invasive breast cancer and explore their correlation with patient outcome following standard neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient has 18 years of age or older at the time of consent.
* The patient has provided pre-treatment tumor samples for WT1 expression screening and gene expression profiling in the context of the NCT01220128 study.
* The patient has a histologically or cytologically confirmed primary invasive breast cancer.
* The patient has provided written informed consent before any new information or new material is provided to the Sponsor.
* The patient is planned to receive, is receiving or has received standard and/or investigational therapy for breast cancer.
* The patient is planned to receive, is receiving or has received standard and/or investigational therapy for breast cancer.

Exclusion Criteria:

Not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who provided a pretreatment tumor sample for Wilms' Tumor 1 (WT1) expression screening in the context of a neoadjuvant interventional study (111172 (WT1-AS15-BRS-001 (NEOADJ)), but who were not included into the active phase of this study.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2011-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The presence of a specific predictive gene expression signature in tumor tissues | At randomization and at definitive surgery which may be up to 30 weeks post randomization.
The presence of immune infiltration in tumor tissues | At randomization and at definitive surgery which may be up to 30 weeks post randomization.
The presence of other candidate biomarkers in tumor tissues | At randomization and at definitive surgery which may be up to 30 weeks post randomization.
The pathological response (complete response or partial response) in the breast. | At definitive surgery which may be up to 30 weeks post randomization.
Disease free interval | Time from definitive surgery to the date of first recurrence of the disease up to maximally 6 years.
Disease free survival | Time from definitive surgery to either the date of first recurrence of the disease or the date of death (whatever the cause), whichever occurs first, up to maximally 6 years.
Overall survival | Time from definitive surgery to the date of death, irrespective of the cause of death. Patients still alive will be censored at the date of the last contact up to maximally 6 years.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- United States (4):
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Amarillo, Texas
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Namur
- Germany (9):
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Kiel, Schleswig-Holstein
- Italy (6):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Aviano (PN), Friuli Venezia Giulia
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Turin, Piedmont
- Russia (2):
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
- United Kingdom (5):
  - GSK Investigational Site, Bournemouth
  - GSK Investigational Site, Derby
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Poole